CLINICAL TRIAL: NCT02608398
Title: The Effect of a Structured Weight-loss Programme on the Metabolic Profiles of Obese and Overweight Children
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 15IC2685
Record Dates: First submitted 2015-08-13; First posted 2015-11-18 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Obesity
Keywords: obesity; weight-loss; metabonomics; gut microbiome
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine and stool samples will be collected from those who consent
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- overweight children at weight-loss camp: This is an observational study there is no intervention. The investigators will carry out metabolic profiling on a cohort of overweight or obese children who are attending a commercial weight loss camp for 2-5 weeks.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — NO intervention by the research group - this is an observational study. urine samples simply collected as children lose weight on their diet and exercise camp

SUMMARY:
Aim:

* The overall aims of this study to look at what changes are seen overweight and obese (very overweight) children, as they get thinner.
* Specifically the investigators are interested in the chemicals and bacteria that children pass in their urine and stool because looking at how these change as it tells us about how their gut and other bodily systems are adapting.

Hypothesis: Metabolic profiling is a useful and accurate tool for observing and monitoring weight loss in children

Study plan:

* To observe this weight loss process in children, the investigators will be attending a commercial weight loss camp called 'MORElife' which takes place every year in Leeds. This camp is attended by children age 8-17years who are overweight or obese, for between two and five weeks. It aims to help them lose weight through a structured diet, exercise, education and support program.
* The investigators plan to, with the consent of the parent and agreement the child ask if they would kindly give us a urine sample at the beginning and end of their time on the camp. For those staying longer than 2 weeks the investigators will also ask for a sample in the middle if possible.
* In addition for those children who consent, the investigators will also ask for a small stool (poo) sample at these same time points although there is no obligation to participate at all in the study and it will not affect their time on the camp whatever they decide.
* Any children who will be attending the MORElife reunion (arranged by the camp at around 10-12 months after) who agree will be asked for a final urine and stool sample to look at the long-term effects.
* Each sample is given a code so as to remain anonymous, frozen and transported to the university laboratory to be analyzed.
* With permission and consent the investigators will also collect some information about the children such as, weight and height from the camp coordinators as well as samples of the diet that they will be fed and example of exercise activities to give a full picture so that results can be as accurate as possible.

DETAILED DESCRIPTION:
STUDY DESIGN

Aims:

1. To identify the effects of a weight-loss programme on the metabolic profiles of obese and overweight children through global profiling of urine, before during and after the intervention.
2. To assess how chemicals (metabolites) in the food eaten by participants compared with those found in their urine through the metabolomic analysis of duplicate meals during the study.

Methodology:

* This will be an observational cohort study type of methodology. A cohort of overweight or obese children who have signed up to a well-known commercial summer weight loss camp (MORElife) will be recruited with parental consent.
* Each child will be attending the MORELife weight loss camp for a minimum of 2 weeks and a maximum of 5 weeks during which time again they are either residential or returning home after 5 pm.
* The programme consists of healthy but hypocaloric balanced meals as well as an exercise programme including a wide range of sports, team games and day trips. Throughout this the children are educated about healthy eating behaviour and choices and given support to achieve a sustained change in lifestyle. At the end of the camp they are followed up for three months by camp support staff via a weekly telephone call to check progress and offer encouragement. During this time and thereafter they can also interact with the support team via social media, email and an interactive web portal.
* Sample collection for metabolic profiling will be in the form of spot urine samples and stool samples from those who wish to and are happy to consent to proved either/both. These will be taken on arrival (Day Zero) prior to commencement of the weight loss programme to give the Control (baseline) sample. Thereafter a 'mid-point' sample will be taken around half way through the camp and a final sample on the day that they leave.
* Associated information for each child such as height, baseline weight on arrival and estimate basal metabolic rate (BMR), and body mass index (BMI) and changes in these parameters through the duration of the camp will be provided to the study by the camp coordinators with parental permission and consent.
* From the samples taken, metabolic profiling of individuals pre- during and post- intervention will be completed using a combination of untargeted and targeted spectroscopic assays including: Nuclear Magnetic Resonance spectroscopy and Mass Spectroscopy profiling of chemicals such as lipids, bile acids, amino acids, bacteria and others found in stool and urine.
* 1-2 meals eaten by the children during the camp will be analysed also by taking a duplicate meal and pureeing it then putting it through similar techniques to the urine and stool samples to compare the chemicals in the food with those excreted from the body.

Participants:

At least 30 male and female children/adolescents aged between 8 and 17 years who are overweight or obese according to classifications for their age. All children in the study will have signed up for the MORElife summer camp 2015 in Leeds, U.K and provided parental consent to take part.

Power calculations:

At the present time there is no data present on the impact of such an intervention in children on the metabolic profile and so such a calculation is not possible, however the numbers that the investigators have chosen reflect other similar studies allowing for a 33.3% drop out rate and the investigators feel confident that they should show representative results.

Health Screening:

Participants will be assessed for suitability to take part in the camp by the organisers of the weight loss camp (MORElife) and so all children who are accepted for entry into the camp will be taken as eligible for this study. The investigators will not be carrying out any separate intervention and are simply collecting samples from them during their time at the camp.

Consent and Participant Information:

Consent forms will be given to the parents of the children prior to beginning the camp as well as information for both parents and children to read before deciding whether they wish to take part. They can contact a member of the research team at any time prior to the study for more information and of course are free to withdraw at any time after agreeing.

Sample collection:

* Each child will be asked to submit a urine sample on day 0 (first day of camp before beginning weight loss programme). Then regular samples will be collected for the duration of their time at the camp with a final one at the reunion around one year later.
* The camp will be asked to provide the investigators with a duplicate lunch and dinner meal to that given to the children so that it can be pureed and prepared for analysis and comparison with the children's metabolic profiles.

Withdrawal Criteria: Children are under no pressure to join the study and can withdraw at any time with no explanation and without their time at Summer camp being affected.

ELIGIBILITY:
Inclusion Criteria:

* All children attending the MORElife Summer Camp with consent

Exclusion Criteria:

* nil

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Overweight or obese children aged between 8-17 years attending the MORElife weight loss Summer Camp
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The effect of a weight-loss programme on the metabolic profile of obese/overweight children (metabolites measured in urine/stool/food using Nuclear Magnetic Resonance Spectrometry and Mass Spectroscopy) | 12 months
  Metabolites detected and compared using Nuclear Magnetic Resonance Spectrometry and Mass Spectroscopy. Using computer software, analysis of these spectra and metabolite identification is carried out and Principal Component Analysis (PCA) completed

CONTACTS AND LOCATIONS:
Overall Officials: Elaine - Holmes, PhD, Study Director — Imperial College London
Locations (1):
- Imperial College London, London, London, United Kingdom